CLINICAL TRIAL: NCT03921164
Title: Non Invasive Pressure -Volume Loop (PVLOOP) With 3D Echocardiography and Arterial Tonometry
Brief Title: Non Invasive Use of Pressure-Volume Loop in the Operating Room
Acronym: LOOPING
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); M3DISIM (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180410; 2018-A02737-48 (Other: IDRCB)
Record Dates: First submitted 2019-04-01; First posted 2019-04-19 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Radiography; Interventional
Keywords: Cardiac after-load; Pressure volume loop; Perioperative risk

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients scheduled for a neuroradiology procedure: Interventional neuroradiology procedure under general anesthesia requiring a continuous monitoring of mean arterial pressure and cardiac output, including electrocardiogram, pulsated oxygen saturation, endtidal CO2, respiratory rate, tidal volume and monitoring of neuromuscular function. In addition, for all patients, data from trans-oesophageal Doppler, trans-thoracic echocardiography (TTE) and hemodynamic data are collected at the end of the procedure. During catheter withdrawal, pressure waveforms are recorded in the descending thoracic aorta just in front of the esophageal Doppler probe.
  Interventions: Procedure: Trans-oesophageal Doppler; Procedure: Trans-thoracic echocardiography; Procedure: Applanation tonometry

INTERVENTIONS:
Procedure: Trans-oesophageal Doppler — As required by the standard of care of the interventional neuroradiology procedure, the neuroradiologist also cannulates the femoral artery. At the end of the procedure, during catheter withdrawal, pressure waveforms are recorded in the descending thoracic aorta just in front of the esophageal Doppler probe.
  Descending aortic velocity is measured with a transesophageal Doppler CardioQ-ODM+ (Deltex Medical, Chichester, UK) in order to construct the VP Loop in descending thoracic aorta.
Procedure: Trans-thoracic echocardiography — Estimation of ventricular diastolic pressure by measuring mitral and aortic flow gradients by echocardiography (EPIQ G7 Philips© or similar) Determination of left ventricular volumes during the cardiac cycle by echocardiography (3D EPIQ G7 Philips© or similar).
  Other Names: TTE
Procedure: Applanation tonometry — Measurements using the SphygmoCor radial tonometer (AtCor Medical, Pty Ltd, Sydney, Australia), the most widely used tonometer in clinical research for non-invasive central pressure measurement and pulse wave analysis. The central blood pressure is then estimated using a validated radial-aortic transfer function.
  The tonometer requires prior calibration by mean (MAP) and diastolic (PAD) blood pressure measured with the conventional brachial cuff as validated in the literature.

SUMMARY:
In patients under general anesthesia, the prevention of intraoperative hypotension to maintain blood pressure (BP) close to the initial blood pressure, i.e. before anesthesia, is essential to reduce the risk of death and improve surgical outcomes. Vasoactive agents are commonly used to correct this hypotension (Phenylephrine Ephedrine Noradrenaline). These three vasoconstrictors have specific effects on the afterload of the heart and can impair its function. The analysis of the left ventricular pressure-volume curve (PV Loop) allows continuous information on the post-charge state of the left ventricle and the changes induced by the vasoconstrictors to be observed. However, the investigators currently have no way of monitoring these effects. In clinical practice if these loops are obtained non-invasively they can be used in the evaluation of cardiac function of at-risk patients in perioperative and also in intensive care to allow therapeutic adaptation.

DETAILED DESCRIPTION:
Investigators have conducted several studies on the differential effects of different vasopressors used in general anesthesia to correct sympatholysis-induced hypotension occurring under anesthetic drugs and after eliminating hypovolemia or overdose in anesthetics.

In a pilot study investigators described a method for analyzing Velocity-Pressure interactions to monitor ventricular afterload in the operating room with the construction of Velocity-Pressure aortic loops (VP Loop).

These loops were constructed from an aortic velocity signal measured by esophageal Doppler and aortic blood pressure signal from a femoral catheter. The Global Afterload Angle (GALA) measured on the loop were then higher in patients at cardiovascular risk (RCV+) at 68 ± 6° compared to 41 ± 15° in patients (RCV-) (p<0.001). In addition, GALA variations were associated with variations in the three components of ventricular afterload: compliance, resistance and waves reflection. Finally, under the effect of vasopressors, there was a modification in the shape of the VP Loop and the value of GALA, showing GALA as a reliable marker potential for ventricular afterload in patients under general anesthesia.

In order to develop a totally non-invasive method that would produce a pressure velocity curve, the investigators propose to combine an estimation of aortic pressure by a tonometry method and an estimation of ventricular volumes by three-dimensional echocardiography.

The main objective of this study is then to compare VP Loop parameters obtained non-invasively to VP loop obtained invasively according to patient cardiovascular risk factors.

Cardiac afterload can be schematically defined by the combination of three components: peripheral vascular resistance (PVR), total arterial compliance (Ctot) and aortic wave reflections (WR). WR could be assessed by pulse wave pressure analysis with the augmentation index (Aix) or after pulse wave pressure separation into a forward and backward wave with the wave reflection index (WRi) or the wave reflection area (WRa).

Invasive Aortic pressure measurements: As required by the standard of care of the interventional neuroradiology procedure, the neuroradiologist also cannulated the femoral artery. At the end of the procedure, during catheter withdrawal, pressure waveforms are recorded in the descending thoracic aorta just in front of the esophageal Doppler probe.

Descending aortic velocity is measured with a transesophageal Doppler CardioQ-ODM+ monitor (Deltex Medical, Chichester, UK) in order to construct the VP Loop in descending thoracic aorta.

Non-invasive Non-invasive Aortic velocity recording VP Loop in aorta is measured in the flushing chamber of the left ventricle from the apical five chamber view by trans-thoracic echocardiography (TTE) (Philips, EPIQ 7).

Estimation of ventricular diastolic pressure by measuring mitral and aortic flow gradients by echocardiography (EPIQ G7 Philips© or similar) Determination of left ventricular volumes during the cardiac cycle by echocardiography (3D EPIQ G7 Philips© or similar).

Non-invasive central pressure measurement by an arterial tonometer reconstructing the central aortic curve (ShygmoCor, AtCor©) The SphygmoCor radial tonometer (AtCor Medical, Pty Ltd, Sydney, Australia) is the most widely used tonometer in clinical research for non-invasive central pressure measurement and pulse wave analysis. The central blood pressure is then estimated using a validated radial-aortic transfer function.

The tonometer requires prior calibration by mean (MAP) and diastolic (PAD) blood pressure measured with the conventional brachial cuff as validated in the literature.

VP Loop construction Digitalization of pressure and velocity signals are performed with the IntelliVue MP60 monitor (Philips, Eindhoven, The Netherlands) at a sampling frequency of 125 Hz and saved using ixTrend software (IXELLENCE, Wildau, Germany) on a computer. Briefly, the velocity coordinates is plotted on the x axis and the pressure coordinates on the y axis. The investigators characterize the VP Loop by 4 points (A, B, C, D), allowing us to identify 3 angles: Alpha, Beta and GALA.

The goal of this study is to compare these parameters of cardiac after load obtained non-invasively with the same parameters invasively obtained.

Experimental design: This is a single-center, interventional, category II prospective study (minimal risks and constraints)

Population concerned: Patients will be included if their perioperative risk required a continuous monitoring of mean arterial pressure (MAP) and cardiac output (CO). The study involves major patients under general anesthesia in interventional neuroradiology.

Research Proceedings For all patients, data from trans-esophageal Doppler, trans-thoracic echocardiography (TTE) and hemodynamic data are collected at the end of the procedure. During catheter withdrawal, pressure waveforms are recorded in the descending thoracic aorta just in front of the esophageal Doppler probe. All data from monitoring are connected to the main monitor.

Individual benefit: There is no benefit for the patient

Collective benefit: Targeting mean arterial pressure (MAP) with boluses of selective peripheral vasopressors (without positive inotropic or chronotropic effects) could have deleterious effects on cardiac output. Thus, it seems important to use a combined analysis of MAP and CO with low invasive methods to estimate the Afterload-related cardiac performance (ACP) in surgical patients considered with "high cardiovascular risk".

Risks and minimal constraints added by the research:

No added risk. Patients are included if their perioperative risk required a continuous monitoring of MAP and CO. The standard of care for the interventional neuroradiology procedure needs a catheterization of the femoral artery using the Seldinger technique and insertion of a catheter. All the other ones measures are obtained non-invasively. Patients are assigned to one of two groups according to their risk of increased arterial stiffness as reported in cardiological publications. The criteria investigators used are as follows: age > 50 years old as a major criterion 20 and cardio-vascular risk factors (history of congestive heart failure, history of cardiovascular event, current smoking, diabetes mellitus, dyslipidemia, and arterial hypertension) as minor criteria. Patients were classified into the high risk group (Hi-risk) if they had at least one major criterion or two minor criteria or into the low risk group (Lo-risk) if they presented with no or one minor criterion. During their interventional neuroradiology procedure, all patients' routine monitoring will consist of electrocardiogram, pulsated oxygen saturation, endtidal carbon dioxide (CO2), respiratory rate, tidal volume and monitoring of neuromuscular function.

For all patients whatever the comorbidities, anesthesia induction will be performed using a target-controlled infusion (Orchestra® Base Primea Fresenius Kabi France). According to our standard of care, intra-operative episodes of hypotension (mean arterial pressure (MAP) < 65 mmHg or < 80% baseline) are treated by Norepinephrine bolus of 10 µg. For all patients, data from trans-esophageal Doppler, trans-thoracic echocardiography (TTE) and hemodynamic data are collected at the end of the procedure.

Number of selected subjects Selection of patients up to 55 analyzable patients Number of centers: 1 Research center Agenda inclusion period: 12 months duration of participation (treatment + follow-up): duration of the interventional neuroradiology procedure: 1 day Total duration: 12 months Number of planned inclusions by center and month: 2-3 Number of subjects required: 55

Statistics: Continuous data are expressed in median [interquartile] and qualitative data in n (%). The risk α has been set at 5%. The categorical variables will be compared by Mann-Whitney test and the continuous variables by Wilcoxon test.

The concordance between the two methods will be evaluated by the intra-class correlation coefficient as well as by the Bland-Altman representation (with determination of bias and approval limits) for the various parameters of interest.

Selection of patients until 55 analyzable patients is obtained (signal quality obtained and possible analysis). The estimate of the number of subjects to be included is based on the main evaluation criterion, the intra-class correlation coefficient. Thus, to highlight, an intra-class correlation coefficient of 0.9 with a confidence interval of 0.1, for an alpha risk of 5%, it is necessary to include 56 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years, scheduled for an elective interventional neuroradiology procedure under general anesthesia requiring a continuous monitoring of mean arterial pressure and cardiac output.

Exclusion Criteria:

* age <18 years
* Patient who has not signed the consent
* Pregnant woman
* Patient under judicial protection
* Patient without affiliation to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for an elective interventional neuroradiology procedure under general anesthesia requiring a continuous monitoring of mean arterial pressure and cardiac output.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Aortic pressure in the descending thoracic aorta in mmHg (PAo) | Duration of the interventional neuroradiology procedure (maximum 1 day)
  For all patients, aortic pressure will be collected at the end of the procedure during catheter withdrawal
Aortic velocity in the descending aorta in cm/s (VAdes.) | Duration of the interventional neuroradiology procedure (maximum 1 day)
  For all patients, aortic descending velocity will be collected at the end of the procedure during catheter withdrawal.
Central pressure by tonometry (CP in mmHg) | Duration of the interventional neuroradiology procedure (maximum 1 day)
  For all patients, central pressure by tonometry will be collected at the end of the procedure.
Ventricular diastolic pressure (VdP in mmHg) | Duration of the interventional neuroradiology procedure (maximum 1 day)
  For all patients, ventricular diastolic pressure by 3D echocardiography will be collected at the end of the procedure.
Left ventricular volume (LVV in mL) | Duration of the interventional neuroradiology procedure (maximum 1 day)
  For all patients, left ventricular volume by 3D echocardiography will be collected at the end of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MATEO, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Fabrice VALLEE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Anesthesiology and Intensive Care, Lariboisière Hospital, Paris, France